CLINICAL TRIAL: NCT05612269
Title: SGLT2 Inhibitors and Reducing the Risk of Cancers Among Diabetics , an Observational Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Amr kamel khalil Ahmed, clinical scientist, Ministry of Health, Saudi Arabia
Other Study IDs: ministry of health
Record Dates: First submitted 2022-10-28; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-10

CONDITIONS: Cancer; Diabetes Mellitus, Type 2; Interleukin 6; SGLT2 Inhibitors
MeSH Terms: conditions — Neoplasms; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: interleukin 6 — follow up of type 2 diabetes with SGLT2 inhibitors like empagliflozin, canagliflozin, and dapagliflozin for measurement of inflammatory factors like interleukin-6, CRP
  Other Names: CRP

SUMMARY:
Since the discovery of SGLT2 inhibitors, there is a great shift in diabetic treatment, so this drug is magic, this drug can reduce the blood sugar level by blocking the reabsorption of glucose in the kidney and increasing glucose excretion the first discovery by Josef von Mering who discovered the glucosuric effect of phlorizin. Phlorizin is the progenitor of contemporary SGLT2 inhibitors, the FDA did not consider the work of Baron Josef von Mering, since he had already discovered acidosis following the administration of phlorizin in 1888.

Now SGLT2 inhibitors are used widely and even for heart failure without diabetes as this drug is useful and with lower risk of death from observational studies The 2008 FDA guidance had a major impact on the cardiovascular (CV) risk assessment of recently approved antidiabetic drugs, many trials were done on SGLT2 inhibitors like the EMPA-REG OUTCOME trial, the CANVAS trial program, MACE these groups have CVS benefits and also renal benefits as regards, we suspect long-term benefits and immunity aspect these groups play an important role in cancer incidence from meta-analysis and systematic review, suggests that SGLT2 inhibition results in a reduction of inflammatory markers like interleukin-6 in animal models, further validating the suggested anti-inflammatory mechanism of action.

DETAILED DESCRIPTION:
The map of treatment of diabetes and obesity was changed dramatically and newer drugs were discovered in the last 10 years for improving the quality of patients and prevent complications and cardiovascular and renal benefits from SGLT2 inhibitors In our study, we will discuss the risk of cancer among diabetics on SGLT2 inhibitors and measurement of inflammatory factors like CRP and interleukin -6 alongside the other investigations the study included 200 adults patients with type 2 diabetes on SGLT2 inhibitors and follow up these patients for one year for the inflammatory factors and risk of cancer among them and this study include patients from 18 years to 70 years having diabetes type 2 male or female, smoker or not smokers, non-diabetic ketoacidosis

ELIGIBILITY:
Inclusion Criteria:

* 18 -70 years male or female diabetics patients smoker or not smokers SGLT-2 inhibitors no history of cancer no severe complications

Exclusion Criteria:

* diabetic ketoacidosis severe diseases pregnant type 1 diabetes

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A study of a group of individuals having diabetes type 2 above 18 years taking any types of SGLT2 inhibitors like canagliflozin, dapagliflozin, and empagliflozin. similar at the disease stage and no history of any type of cancer we will measure the interleukin 6 and CRP among these patients and follow up for one year for calculating the risk of occurrence of any type of cancer
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Reducing the risk of cancer among Diabetics with SGLT2 inhibitors | 9 month after treatment

SECONDARY OUTCOMES:
measurement of inflammatory factors like interleukin-6 | 9 month after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- ministry of health , First health cluster , Riaydh, Riyadh, N/A (Non-US), Saudi Arabia

IPD SHARING:
Plan to Share IPD: No